CLINICAL TRIAL: NCT02851355
Title: Follow-up Survey of Patients Who Were Treated for Medulloblastoma or Primitive Neuroectodermal Tumors of the Central Nervous in Norway
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Einar Stensvold, M.D, Oslo University Hospital
Other Study IDs: 2015/2362
Record Dates: First submitted 2016-06-22; First posted 2016-08-01 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical follow-up survey of the Norwegian material of paediatric patients who received therapy for medulloblastoma and CNS-PNET from 1974 - 2013 with a focus on quality of life, education, work, family and children, delayed effects of tumour disease and treatment, endocrine evaluation, existence of auditory neuropathy, and neuropsychological testing.

ELIGIBILITY:
Inclusion Criteria:

* Whose who has been treated for medulloblastoma og CNS-PNET between 1974 and 2013

Exclusion Criteria:

* Other brain tumours

Ages: 5 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Those children and adolescents who were younger than 18 years of age and who recived treatement for medulloblastoma or CNS-PNET in southern part of Norway between 1974 and 2013.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
SF 36 for those older than 18 years | 1 year
  Questionnaire
PedsQL for those younger than 18 years | 1 year
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Einar Stensvold, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No